CLINICAL TRIAL: NCT06140056
Title: Transpulmonary Pressure During Volume Controlled Mechanical Ventilation Versus Airway Pressure Release Ventilation for Hypoxic Respiratory Failure - a Randomized Feasibility Study
Brief Title: Two Modes of Mechanical Ventilation for Intensive Care Patients With Low Blood Oxygen Due to Breathing Difficulties
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated early due to slower than expected recruitment and limited resources for further enrollment.
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Theis S. Itenov, Sponsor, University Hospital Bispebjerg and Frederiksberg
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: H-23050947
Record Dates: First submitted 2023-10-02; First posted 2023-11-18 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Hypoxic Respiratory Failure; Ventilators, Mechanical
Keywords: Transpulmonary pressure; Airway pressure release ventilation; Volumen controlled mechanical ventilation; Esophageal pressure; Esophageal manometry
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Duration: 3 hours
  Interventions: Other: Volumen controlled mechanical ventilation
- Intervention (Experimental): Duration: 3 hours
  Interventions: Other: Airway pressure release ventilation

INTERVENTIONS:
Other: Airway pressure release ventilation — Mechanical ventilation mode
  Arms: Intervention
Other: Volumen controlled mechanical ventilation — Mechanical ventilation mode
  Arms: Control

SUMMARY:
The study examines individuals admitted to the intensive care unit due to breathing difficulties resulting in not getting enough oxygen into their bodies. These patient will receive mechanical ventilation and this study aims to determine how the pressure inside the lungs changes when using two different modes of mechanical ventilation. The goal is to improve management and care of breathing difficulties by gaining insight into changes in lung pressure during mechanical ventilation, as well as comparing the effectiveness of the two ventilator modes.

DETAILED DESCRIPTION:
As hypoxic respiratory failure is an acute condition, this trial will enrol temporarily incompetent patients and obtain consent from the patient's next of kin and an independent medical doctor (trial guardian) as soon as possible after enrolment.

When included in the study, patients will be randomized 1:1 centrally in the RedCap system, using a computer-generated concealed assignment sequence, with permuted blocks of varying sizes, to start with either the intervention (APRV) followed by control (volume controlled mechanical ventilation) or control followed by intervention.

Esophageal manometry will be used as a surrogate to measure the transpulmonary pressure. Arterial blood gasses, blood samples and lung ultrasound will be used to investigate oxygenation, ventilation and aeration.

Treatment targets for both groups during the study are pH >7.20, saturation ≥ 88% and PaO2 ≥ 8.0 kPa, with FiO2 titrated as low as possible while complying to the oxygenation targets (PaO2 and saturation).

Both arms start with an 'adjustment phase' where the ventilator is adjusted so the respiratory values are within the targets. The intervention adjustment phase is at least 30 minutes. The adjustments will follow standardized protocols.

When the respiratory values are within range, the 'observation period begins' and no changes are made to the ventilator for 3 hours, unless it is necessary to achieve ventilatory treatment targets or deemed necessary by the treating physician. During the trial, the patient must be positioned in a supine position with the headboard elevated 0-30 degrees.

After the first 'observation period', the patient is switched to the opposite ventilation mode and will go through an 'adjustment phase' and 'observation period' again.

Once a patient regains competence, they will be provided with both written and oral information regarding the trial

By comparing volume controlled mechanical ventilation and APRV and their transpulmonary pressures, valuable insight can be gained regarding optimal ventilation strategy for patients with hypoxic respiratory failure. Understanding how various ventilation modes influence transpulmonary pressure and their potential effects on respiratory mechanics can potentially inform designs of trials with individualized respiratory care.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the ICU
* Invasive mechanical ventilation with FiO2 ≥ 50% OR PaO2-to-FiO2 ratio <20 kPa, including PEEP 3 5 cmH20 for at least 6 hours

Exclusion Criteria:

* Meeting inclusion criteria for more than 24 hours
* Severe bronchospasm, defined as warranting treatment aimed at reversing this i.e. inhalation of anticholinergic or bronchodilator beyond what the patient normally use
* Emphysema where treating physician judges the patient at increased risk for pneumothorax from APRV
* Restrictive lung disease defined as a pre-admission diagnosis of restrictive lung disease
* Undrained pneumothorax
* Hemodynamic instability defined as more than 0.20 microgram/kg/min of norepinephrine or any dose of adrenaline infusion to maintain MAP ≥ 65 mmHg
* Age < 18 years
* Patients who have received APRV previously during the current ICU admission
* Patients in prone position within the last 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2025-08-03 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Median peak transpulmonary pressure | During the observation period; 1-6 hours after randomization
  Measured with esophageal manometry in cmH20.

SECONDARY OUTCOMES:
Proportion of patients with peak transpulmonary pressure > 12 cmH2O | During observation period; 1-6 hours after randomization
  Measured with esophageal manometry
Change in peak transpulmonary pressure in cmH20 | During observation period; 1-6 hours after randomization
  Measured with esophageal manometry. Calculated as beginning - end of observation period
Fluctuations in transpulmonary pressure in cmH20 | During observation period; 1-6 hours after randomization
  Measured with esophageal manometry. Difference between peak and nadir transpulmonary pressure during respiratory cycle
Change in fluctuations of transpulmonary pressure in cmH20 | During observation period; 1-6 hours after randomization
  Measured with esophageal manometry. Calculated as beginning - end of observation period.
Nadir PaO2-to-FiO2 ratio | During observation period; 1-6 hours after randomization
  Calculated by PaO2/FiO2. PaO2 from arterial blood gasses and FiO2 from ventilator setting
Peak FiO2 in % | During observation period; 1-6 hours after randomization
  FiO2 from ventilator settings
Peak PaCO2 in kPa | During observation period; 1-6 hours after randomization
  PaCO2 from arterial blood gasses
Nadir pH | During observation period; 1-6 hours after randomization
  pH from arterial blood gasses
Lung ultrasound aeration according to LUS | During observation period; 1-6 hours after randomization
  Evaluating lung aeration by Lung Ultrasound Score

OTHER OUTCOMES:
Proportion of patients unable to tolerate observation period without increasing ventilator settings | During observation period; 1-6 hours after randomization
  Defined as measures aimed at increasing either oxygenation or ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Theis S Itenov, MD, PhD, Principal Investigator — University Hospital Bispebjerg and Frederiksberg
Locations (2):
- Denmark (2):
  - Bispebjerg Hospital, Copenhagen
  - Hvidovre Hospital, Hvidovre

IPD SHARING:
Plan to Share IPD: Yes
All data will be owned by the steering committee. De-identified data will be made available 1 year after the primary publication of the outcome data. The statistical code will be submitted as an appendix to primary publication.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: A year after publication of the primary outcome data
Access Criteria: By written request to the steering committee. The sharing of data must be subject to a written agreement between the Capital Region of Denmark and receiver, and in accordance with data regulations. The steering committe will ensure that this.